CLINICAL TRIAL: NCT05283824
Title: Comparison of 3 Techniques for Blood Pressure Measurements During Interventional Neuroradiology Procedures
Acronym: NEXFIN-NRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: NEXFIN-NRI( 29BRC21.0268)
Record Dates: First submitted 2022-02-07; First posted 2022-03-17 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some observational studies demonstrated that hypotension was associated with post-operative morbidity. During neuroradiological procedures, cerebral perfusion pressure should be cautiously maintained and hypertension should also be avoided. So, a precise arterial pressure measurement is needed during this procedures. A continuous monitoring of arterial pressure needed the placement of an arterial catheter in radial artery. The placement of this catheter might be long, difficult and incompatible with emergency neuroradiological procedure (such as thrombectomy). Then, this invasive technique is associated with several minor and major side effects such as: pain, infection, thrombosis, hematoma.

The Clearsight®, commercialized by Edwards Life Science Company®, is a non invasive device which mesure continuously arterial pressure with Volume-Clamp method. In operating room, some studies found a good accuracy between Clearsight® and other invasive monitoring system. There is no description of the use of Clearsight® during neuroradiological procedures.

The investigators hypothesized that Clearsight® measurement of arterial pressure are concordant with arterial pressure measure with the placement of an arterial catheter. The investigators also plan to evaluate accuracy of intermittent non invasive pressure measurement with traditional cuff.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age > 18 years old)
* Elective or emergent neuroradiological procedure under general or local anesthesia for : Endovascular treatment of cerebral aneurysms / arteriovenous malformation, Thrombectomy, Arteriography, transluminal balloon angioplasty for vasospasm
* Placement of arterial catheter for the measurement of continuous arterial pressure

Exclusion Criteria:

* Contraindication of placement of arterial catheter or digital cuff (Clearsight) such as: Reynaud syndrome, Buerger syndrome
* Pregnant women
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, admitted in operating room elective or emergent neuroradiological procedure
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Systolic arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of systolic arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (Clearsight©)
Diastolic arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of diastolic arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (Clearsight©)
Mean arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of mean arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (Clearsight©)

SECONDARY OUTCOMES:
Systolic arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of systolic arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (classical harm cuff)
Diastolic arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of diastolic arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (classical harm cuff)
Mean arterial blood pressure (mmHg) | During neuroradiological procedure
  The main objective of this study is to evaluate concordance of mean arterial pressure pressure (in mmHg) measurement between invasive (arterial catheter) and non invasive technique (classical harm cuff)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier CHAPALAIN, MD, Principal Investigator — Department of Anesthesiology and Surgical ICU, Brest University Hospital
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Kim SH, Lilot M, Sidhu KS, Rinehart J, Yu Z, Canales C, Cannesson M. Accuracy and precision of continuous noninvasive arterial pressure monitoring compared with invasive arterial pressure: a systematic review and meta-analysis. Anesthesiology. 2014 May;120(5):1080-97. doi: 10.1097/ALN.0000000000000226. PMID 24637618
- [Result] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Result] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Result] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Result] Hofhuizen C, Lansdorp B, van der Hoeven JG, Scheffer GJ, Lemson J. Validation of noninvasive pulse contour cardiac output using finger arterial pressure in cardiac surgery patients requiring fluid therapy. J Crit Care. 2014 Feb;29(1):161-5. doi: 10.1016/j.jcrc.2013.09.005. PMID 24475498
- [Result] Chen G, Meng L, Alexander B, Tran NP, Kain ZN, Cannesson M. Comparison of noninvasive cardiac output measurements using the Nexfin monitoring device and the esophageal Doppler. J Clin Anesth. 2012 Jun;24(4):275-83. doi: 10.1016/j.jclinane.2011.08.014. PMID 22608581
- [Derived] Chapalain X, Morvan T, Gentric JC, Subileau A, Jacob C, Cadic A, Caillard A, Huet O. Continuous non-invasive vs. invasive arterial blood pressure monitoring during neuroradiological procedure: a comparative, prospective, monocentric, observational study. Perioper Med (Lond). 2024 Jul 22;13(1):77. doi: 10.1186/s13741-024-00442-3. PMID 39034414
- See also: Volume-Clamp Method — https://www.atlantis-press.com/proceedings/meic-15/19790